# Statistical Analysis Plan

A Phase 3 Multi-Center, Open Label Study Evaluating the Long Term Safety of SB204 Once Daily in the Treatment of Acne Vulgaris

> Novan, Inc. 4105 Hopson Road Morrisville, NC 27560

Author(s): Melissa Hays

Document Status: Final

Version Date: Version 1.0 12Apr2017

Novan, Inc.

## Contents

| A | bbrev | iations | 3 |
|---|-------|------------------------------------------|-----|
| 1 | ] | Introduction | . 4 |
| 2 | 5 | Study Objectives | 4 |
| | 2.1 | Safety Endpoints | . 4 |
| | 2.2 | Tolerability Endpoints | |
| | 2.3 | Extent of Exposure | |
| | 2.4 | Efficacy Endpoints | . 4 |
| 3 | 9 | Study Design | . 4 |
| | 3.1 | Study Design | 4 |
| | 3.2 | Study Treatment | . 5 |
| | 3.3 | Study Schedule | . 6 |
| | 3.4 | Concomitant Medication | 7 |
| | 3.5 | Populations | . 7 |
| | 3.5.1 | Safety Population | . 7 |
| | 3.6 | Sample Size | . 7 |
| 4 | 5 | Statistical Methodology | . 8 |
| | 4.1 | Planned Analyses | . 8 |
| | 4.2 | Disposition of Subjects | . 8 |
| | 4.3 | Baseline and Demographic Characteristics | . 8 |
| | 4.4 | Extent and Duration of Exposure | . 8 |
| | 4.5 | Safety | . 9 |
| | 4.5.1 | Adverse Events | . 9 |
| | 4.5.2 | Prior and Concomitant Medications | 10 |
| | 4.5.3 | Physical Examination | 10 |
| | 4.5.4 | Vital Signs | |
| | 4.5.5 | Urine Pregnancy Tests | |
| | 4.6 | Tolerability | |
| | 4.7 | Efficacy Analysis | |
| | 4.8 | Deviations from SAP | 11 |

# **Abbreviations**

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| AE | Adverse Event |
| ATC | Anatomical and Therapeutic Class |
| ET | Early Termination |
| g | gram |
| IRB | Institutional Review Board |
| LTS | Long-Term Safety |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NOVAN | Novan, Inc. |
| OCP | Oral Contraceptive Pill |
| PT | Preferred Term |
| SAE | Serious Adverse Event |
| SAF | Safety Population |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis Software |
| SOC | System Organ Class |
| TEAE | Treatment Emergent Adverse Events |
| UPT | Urine Pregnancy Test |
| WHO | World Health Organization |
| WOCBP | Women of Child-Bearing Potential |

### 1 Introduction

This document presents the statistical analysis plan (SAP) for Novan Inc., Protocol No. NI-AC303: A Phase 3 Multi-Center, Open Label Study Evaluating the Long Term Safety of SB204 Once Daily in the Treatment of Acne Vulgaris.

The SAP provides the detailed description of the planned statistical analysis of data from protocol NI-AC303.

## 2 Study Objectives

The primary objective of this study is to evaluate the safety of SB204 4% once daily in subjects with acne vulgaris for up to 40 weeks of treatment. The Week 12 visit from the pivotal studies (NI-AC301 and NI-AC302) will serve as the Baseline Visit for this study.

#### 2.1 Safety Endpoints

Safety endpoints will include adverse events, changes in physical examination and changes in vital sign measurements. Any clinically significant changes noted during the physical exam as well as from the vital sign measurements will be recorded as adverse events and included in the comparison. Urine pregnancy tests in women of child-bearing potential will be conducted at each visit.

### 2.2 Tolerability Endpoints

The cutaneous tolerability assessments include the investigator's assessment of erythema, scaling, dryness, and the subject's report of pruritus and burning/stinging based on the preceding 24 hours.

### 2.3 Extent of Exposure

Duration, days of, and extent of exposure for each subject will be determined based on the stop and start dates of use of SB204, the total number of days of study drug application, and the areas treated (face, upper back, upper chest, and shoulders).

### 2.4 Efficacy Endpoints

Efficacy endpoints will include absolute and percent change in inflammatory and non-inflammatory facial area lesion counts from baseline at each study visit.

# 3 Study Design

### 3.1 Study Design

This is a multi-center, open label long-term safety (LTS) study to be conducted in approximately 600 subjects with acne vulgaris. Subjects will be enrolled into the study from approximately 100

sites in North America. Subjects eligible to enroll in this study will have completed one of the Phase 3 pivotal studies with SB204, NI-AC301 or NI-AC302, and meet study inclusion and exclusion criteria.

Subjects who satisfy the entry criteria at the Baseline visit will be enrolled to receive open-label SB204. Investigational drug will be delivered from a double barrel single pump dispenser. The pump dispenses product (NVN1000 Gel and a hydrogel) from two chambers which will be mixed together quickly (about 5 seconds) by the subject and applied once daily to the acne affected areas identified by the Investigator. Areas that could be treated include the face, upper chest, upper back and shoulders. No other acne treatments will be permitted during the study.

Subjects will return for post-baseline evaluation at Weeks 4, 12, 24, 36 and 40/ET.

#### 3.2 Study Treatment

The amount of SB204 per application will vary depending on the areas to be treated as shown in Table 1 below. Subjects are allowed to specify 'Other'. If the other specification is jaw or neckline, it is assumed that the same pump stroke used to apply drug to face is being used for the jaw and/or neckline application. One pump stroke will likely be used for each application area. For example, application to the face, upper back and upper chest will require up to 2.7 g (three (3) pump strokes).

**Table 1: Dosing Amount by Area** 

| Area (BSA) | Number of Pump Strokes | Amount of Product |
|---|---|---|
| Face, including jaw line and or neck if indicated | 1 | 0.9 g |
| Upper Back | 1 | 0.9 g |
| Upper Chest | 1 | 0.9 g |
| Shoulders | 1 | 0.9 g |

### 3.3 Study Schedule

Study visits should occur at approximately the same time of day throughout the study.

| PROCEDURES | Visit 1 <sup>1</sup> Baseline (Day 0) | Visit 2 <sup>3</sup><br>Week 4<br>±5 days<br>(Day 28) | Visit 3<br>Week 12<br>±7 days<br>(Day 84) | Visit 4<br>Week 24<br>±7 days<br>(Day 168) | Visit 5<br>Week 36<br>±7 days<br>(Day 252) | Visit 6 <sup>4</sup><br>Week 40/ET<br>±7 days<br>(Day 280) |
|---|---|---|---|---|---|---|
| Informed | X | | | | | |
| Consent/Assent | | | | | | |
| Demographics | $X^2$ | | | | | |
| Medical History | X | | | | | |
| Medication History | X | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | |
| Brief Physical<br>Examination | $X^2$ | | | | | X |
| Urine Pregnancy Test (all WOCBP) | $X^2$ | X | X | X | X | X |
| Blood Pressure and<br>Pulse | $X^2$ | X | X | X | X | X |
| Lesion Counts | $X^2$ | X | X | X | X | X |
| Cutaneous Tolerability Evaluation | $X^2$ | X | X | X | X | X |
| Instruct on Study Drug Application and Provide Subject Instructions | X | | | | | |
| Record application areas since last visit | | X | X | X | X | X |
| Study Drug Dispensed/Retraining on mixing and application | X | X | X | X | X | |
| Study Drug Collected | | X | X | X | X | X |
| Subject Study Drug Use<br>Reviewed | | X | X | X | X | X |
| Concomitant<br>Medications | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X |

<sup>&</sup>lt;sup>1</sup>Data for the Baseline Visit for this study will be the Week 12 data from the Phase 3 pivotal study for completing, eligible subjects.

<sup>&</sup>lt;sup>2</sup>Demographics and assessments from the Week 12 visit from the preceding Phase 3 study including the physical examination, blood pressure and pulse, UPT, tolerability, and lesion counts do not need to be repeated.

<sup>&</sup>lt;sup>3</sup>All visit dates are in reference to Baseline, e.g., Visit 2 occurs four weeks (28 days) after Baseline visit.

<sup>&</sup>lt;sup>4</sup>All Week 40 procedures should be completed for subjects who prematurely discontinue, if possible.

#### 3.4 Concomitant Medication

Subjects will be permitted to apply non-comedogenic moisturizer or sunscreen on an as-needed basis. Moisturizer must not contain antibacterials and the subject must not change moisturizer and/or sunscreen used during the course of the study. If used, moisturizers and sunscreen must be applied at least 30 minutes after study drug application.

Subjects must not have used anti-acne treatments including topical or systemic antibiotics or retinoids (as described in Section 3.7.3 of the protocol) prior to Baseline. These medications are also prohibited during the trial. Short term courses of antibiotics ( $\leq$  14 days) for non-acne related illnesses and inhaled or intranasal steroids are permitted during the trial.

Subjects may not be concurrently on drugs associated with exacerbating acne vulgaris (see Appendix 16.1 of the protocol). Subjects must not participate in a different interventional research study during the study period.

Any medication/therapy used by the subject following first application of study product will be considered a concomitant medication/therapy (e.g., aspirin, acetaminophen, birth control pills, vitamins, etc.). Every attempt should be made to keep concomitant medication/therapy dosing constant during the study. Any change to concomitant medications/therapies should be noted on the subject's study record and in the study database. When applicable, an AE should be completed for any subject starting a concomitant medication/therapy after enrollment into the study.

#### 3.5 Populations

#### 3.5.1 Safety Population

The safety population (SAF) will include all subjects that have received at least one dose of SB204. For the summaries, we are defining two subject categories, based on the subject's status at the start of the LTS:

- SB204 Experienced: subjects allocated to SB204 in the previous study
- SB204 Naïve: subjects allocated to vehicle in the previous study

### 3.6 Sample Size

The main objective of this study is to evaluate the long term safety of SB204, therefore, no sample size or power calculations were performed.

# 4 Statistical Methodology

#### 4.1 Planned Analyses

All statistical processing will be performed using statistical analysis software (SAS®) unless otherwise stated. Safety analyses will be performed using the safety population.

Continuous data will be summarized with sample size (N), mean, median, standard deviation, minimum and maximum. Categorical data will be summarized with N, frequency counts, and percentages, based on N.

#### 4.2 Disposition of Subjects

The number of subjects in the Safety Population, who completed the study and the reasons for any premature discontinuation from the study, will be presented. Listings will indicate whether subjects met all inclusion and exclusion criteria, and, if not, which criteria were not met.

A summary and a listing of protocol deviations will be presented.

### 4.3 Baseline and Demographic Characteristics

Subject baseline and demographic characteristics, including age, race, ethnicity, and gender, will be summarized, as well as which previous Novan study the subject was enrolled in (NI-AC301 or NI-AC302) and previous treatment assignment (SB204 or Vehicle).

For female subjects the following summaries will be included: child-bearing potential, contraceptive use at baseline. Medical history will be summarized for each treatment group by SOC and PT and presented in listings. Adverse events ongoing at end of pivotal study will be carried forward to this study, will not be considered treatment-emergent for this study, and will be summarized separately by SOC, PT, and relatedness.

### 4.4 Extent and Duration of Exposure

Summaries of the duration of exposure, days of exposure, and extent of exposure (calculated total grams) to study drug will be presented, overall and by whether previously randomized to SB204 (SB204 experienced) or randomized to Vehicle (SB204 naïve). This information plus study drug management details will be listed as well. All exposure endpoints will take into account whether the subject received SB204 in the previous study (NI-AC301 or NI-AC302).

Duration of exposure will be defined as:

Date of Last Drug Administration – Date of First Drug Administration + 1 day

Where date of first drug administration is the date of first treatment in the previous pivotal study for subjects randomized to SB204 in the previous study, and date of first dose in the LTS for subjects randomized to vehicle in the previous study.

Days of exposure will be defined as the total number of days that the subject reported taking study medication, and includes the days of exposure to SB204 in the previous study (NI-AC301 or NI-AC302) if applicable.

Extent of exposure will be based on the number of areas treated (face, upper back, and/or upper chest/shoulders, and any other areas reported) and the number of days with treatment. For subjects randomized to SB204 in the previous studies, drug was only applied to the face so for the days of exposure from the previous studies, it will be assumed that there is only one area of application, i.e. the face.

Each application is equal to 0.9 g. Extent of exposure is estimated as the sum of application areas (face only=1, face and chest=2, etc.) times the number of days of application to those areas times 0.9g. For example, a subject who applies 200 applications to the face only will have extent of exposure = 180g, while a subject who applies 100 applications to the face and 50 applications to the upper back will have extent of exposure = 135 g. The maximum extent of exposure would be: [0.9 grams x number of days on treatment in previous study] + [0.9 grams x 4 areas x number of LTS days on treatment]. Most subjects will have less exposure than this, so extent of exposure will be categorized logically depending on actual distribution of subjects. Initially, quartiles will considered.

#### 4.5 Safety

#### 4.5.1 Adverse Events

All AEs that occur during the study or continue after enrollment into this study will be recorded and classified on the basis of Medical Dictionary for Regulatory Activities (MedDRA) terminology version 18.1. Adverse events ongoing at end of the pivotal study will be carried forward to this study, will not be considered treatment-emergent for this study, and will be summarized separately by SOC, PT, and relatedness. Treatment-emergent AEs (TEAEs) will be defined as AEs reported on or after the first day of enrollment in this long term safety study.

All information pertaining to an AE noted during the study will be listed by subject, detailing verbatim term given by the Investigator or designee, preferred term, system organ class (SOC), onset date, resolution date, severity, seriousness, action taken, outcome, and drug relatedness. The event onset will also be shown relative (in number of days) to date of first dose in this study.

Treatment-emergent AEs will be summarized by the number of subjects reporting a TEAE, SOC, preferred term, severity, relationship to study drug (causality), and seriousness. When summarizing AEs by severity and relationship, each subject will be counted only once, within a system organ class or a preferred term, by using the event with the highest severity and greatest relationship within each classification.

Serious AEs will be summarized by severity, and relationship to study drug, and individual SAEs will be listed by subject. In addition, a list of subjects who prematurely discontinue study drug due to an AE, had AEs leading to treatment modification, and AEs that resulted in death will be provided.

Adverse events will also be summarized by windows of duration of exposure to study drug to determine if there is a safety signal due to duration of exposure. The windows of exposure will include but are not limited to: 1) within the first 24 hours (i.e. Day 1 of the LTS study), 2) up to 1 month (i.e. 2-30 days), 3) up to 3 months (i.e. 31-90 days), 4) up to 6 months (i.e. 91-180 days) and 5) up to 12 months (i.e. 181-365 days).

Adverse event incidence will also be summarized by the extent of exposure categories (in grams) as described in section 4.4.

#### 4.5.2 Prior and Concomitant Medications

Medications will be mapped to their corresponding thesaurus terms (ATC Class and Preferred Term) according to the World Health Organization (WHO) Drug Dictionary, Version Mar2016. A summary of concomitant medications, sorted by ATC Class 2 and Preferred Term, will be provided. A listing of prior and concomitant medications will be presented, as well a listing of any prohibited medications used during the study.

#### 4.5.3 Physical Examination

The results of the physical exams will be presented in a listing. Clinically significant changes from Baseline will be documented as an AE.

#### 4.5.4 Vital Signs

Blood pressure and pulse will be summarized from Baseline through Week 40/ET. Additionally, change from Baseline in vital signs will be summarized at Week 4, 12, 24, 36, and 40/ET. Clinically significant changes from Baseline will be documented as an AE.

#### 4.5.5 Urine Pregnancy Tests

Urine pregnancy tests results for WOCBP will be presented in data listings by subject.

### 4.6 Tolerability

Distribution and shift in cutaneous tolerability assessments (erythema, scaling, dryness, pruritus, burning/stinging) will be summarized from Baseline to Week 40/ET.

### 4.7 Efficacy Analysis

The facial area inflammatory and non-inflammatory lesion counts will be summarized at each evaluation from Baseline through Week 40/ET. Absolute and percent change in inflammatory and non-inflammatory lesion counts will be summarized at Weeks 4, 12, 24, 36 and 40/ET. The absolute and percent change in inflammatory non-inflammatory lesion counts will also be summarized by prior treatment (SB204 experienced, SB204 naïve).

#### 4.8 Deviations from SAP

Any deviations from the original statistical plan will be described and justified in the final clinical study report.

Protocol: NI-AC303

A Phase 3 Multi-Center, Open Label Study Evaluating the Long Term Safety of SB204 Once Daily in the Treatment of Acne Vulgaris.

Mock Data Displays- Tables Version 1.0 Date: 12Apr2017

Prepared for:
Novan Inc.
4105 Hopson Road
Morrisville, NC 27560

Prepared by:
Chiltern International
4000 CentreGreen Way, Suite 300, Cary, NC, 27513, United States

This document is the confidential information of Novan Inc. It may not be disclosed to parties not associated with the clinical investigation or used for any purpose without the prior written consent of Novan Inc.

#### Contents

| Table 14.1.1.1 Subject Disposition Safety Population | 4 |
|---|---|
| Table 14.1.1.2 Summary of Protocol Deviations Safety Population | 5 |
| Table 14.1.2.1 Demographics Safety Population | 6 |
| Table 14.1.2.2 Child Bearing Potential and Contraceptive Use (Females Only) Safety Population | 7 |
| Table 14.1.3 Medical History by System Organ Class and Preferred Term Safety Population | |
| Table 14.1.4 Adverse Events Ongoing at the Start of the Study by System Organ Class, Preferred Term, and Extent of Exposure Safety Population | 9 |
| Table 14.1.5 Concomitant Medications by WHO Drug Class and WHO Drug Preferred Name Safety Population | 10 |
| Table 14.2.1. Summary of Duration and Extent of Drug Exposure Safety Population | |
| Table 14.2.2.1 Inflammatory Lesion Counts by Study Visit (Face Only) Safety Population | 12 |
| Table 14.2.2.2 Non-Inflammatory Lesion Counts by Study Visit (Face Only) Safety Population | |
| Table 14.2.3.1 Inflammatory Lesion Counts (Face Only) by Prior Treatment and Study Visit Safety Population | 13 |
| Table 14.2.3.2 Non-Inflammatory Lesion Counts (Face Only) by Prior Treatment and Study Visit Safety Population | 13 |
| Table 14.3.1.1 Cutaneous Tolerability Evaluation – Erythema - Summarized by Study Visit (Face Only) Safety Population | 14 |
| Table 14.3.1.2 Cutaneous Tolerability Evaluation – Scaling - Summarized by Study Visit Safety Population | 15 |
| Table 14.3.1.3 Cutaneous Tolerability Evaluation – Dryness - Summarized by Study Visit Safety Population | 15 |
| Table 14.3.1.4 Cutaneous Tolerability Evaluation – Pruritus - Summarized by Study Visit Safety Population | 15 |
| Table 14.3.1.5 Cutaneous Tolerability Evaluation – Burning/Stinging - Summarized by Study Visit Safety Population | |
| Table 14.3.2.1 Shift from Baseline in Cutaneous Tolerability Evaluation – Erythema, by Study Visit (Face Only) Safety Population | 16 |
| Table 14.3.2.2 Shift from Baseline in Cutaneous Tolerability Evaluation – Scaling - Summarized Continuously by Study Visit Safety Population | |
| Table 14.3.2.3 Shift from Baseline in Cutaneous Tolerability Evaluation – Dryness - Summarized Continuously by Study Visit Safety Population | |
| Table 14.3.2.4 Shift from Baseline in Cutaneous Tolerability Evaluation – Pruritus - Summarized Continuously by Study Visit Safety Population | |
| Table 14.3.2.5 Shift from Baseline in Cutaneous Tolerability Evaluation – Burning/Stinging - Summarized Continuously by Study Visit Safety Population | |
| Table 14.3.3.1 Treatment Emergent Adverse Events (TEAE) Overview Safety Population | 18 |
| Table 14.3.3.2.1 Treatment Emergent Adverse Events (TEAE) by System Organ Class, Preferred Term, and Duration of Exposure Safety Population | 19 |
| Table 14.3.3.2.2 Treatment Emergent Adverse Events (TEAE) by System Organ Class, Preferred Term, and Extent of Exposure Safety Population | |
| Table 14.3.3.3.1 Treatment-Related Emergent Adverse Events by System Organ Class, Preferred Term, and Duration of Exposure Safety Population | 21 |
| Table 14.3.3.3.2 Treatment-Related Emergent Adverse Events by System Organ Class, Preferred Term, and Extent of Exposure Safety Population | |
| Table 14.3.3.4.1 Treatment Emergent Adverse Events Leading to Treatment Modification by Duration of Exposure Safety Population | 21 |
| Table 14.3.3.4.2 Treatment Emergent Adverse Events Leading to Treatment Modification by Extent of Exposure Safety Population | 21 |
| Table 14.3.3.5.1 Treatment-Related Treatment Emergent Adverse Events Leading to Treatment Modification by Duration of Exposure Safety Population | |
| Table 14.3.3.5.2 Treatment-Related Treatment Emergent Adverse Events Leading to Treatment Modification by Extent of Exposure Safety Population | |
| Table 14.3.3.6.1 Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug by Duration of Exposure Safety Population | |
| Table 14.3.3.6.2 Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug by Extent of Exposure Safety Population | |
| Table 14.3.3.7.1 Treatment-Related Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug by Duration of Exposure Safety Popular | ation |
| | 21 |
| Table 14.3.3.7.2 Treatment-Related Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug by Extent of Exposure Safety Population | 22 |

Protocol Number: NI-AC303

| Table 14.3.3.8.1 Treatment Emergent Serious Adverse Events by System Organ Class, Preferred Term, and Duration of Exposure Safety Population | 22 |
|---|---|
| Table 14.3.3.8.2 Treatment Emergent Serious Adverse Events by System Organ Class, Preferred Term, and Extent of Exposure Safety Population | 22 |
| Table 14.3.3.9.1 Treatment-Related Treatment Emergent Serious Adverse Events by System Organ Class, Preferred Term, and Duration of Exposur | re Safety |
| Population | 22 |
| Table 14.3.3.9.2 Treatment-Related Treatment Emergent Serious Adverse Events by System Organ Class, Preferred Term, and Extent of Exposur | re Safety |
| Population | 22 |
| Table 14.3.3.10.1 Treatment Emergent Adverse Events Leading to Death by Duration of Exposure Safety Population | 22 |
| Table 14.3.3.10.2 Treatment Emergent Adverse Events Leading to Death by Extent of Exposure Safety Population | 22 |
| Table 14.3.3.11.1 Treatment-Related Treatment Emergent Adverse Events Leading to Death by Duration of Exposure Safety Population | 22 |
| Table 14.3.3.11.2 Treatment-Related Treatment Emergent Adverse Events Leading to Death by Extent of Exposure Safety Population | 22 |
| Table 14.3.3.13 Summary of Treatment Emergent Adverse Events (TEAE) by Highest Severity, System Organ Class and Preferred Term Safety Populat | tion23 |
| Table 14.3.3.14 Summary of Treatment-Related Emergent Adverse Events (TEAE) by Severity, System Organ Class and Preferred Term Safety Population | ion24 |
| Table 14.3.4 Summary of Vital Signs Safety Population | 25 |

Protocol Number: NI-AC303

Table 14.1.1.1
Subject Disposition
Safety Population

| | SB204 |
|------------------------------------------------|-----------|
| | (N=XXX) |
| SAF Population | xx (xx.x) |
| Treatment-naïve at enrollment | xx (xx.x) |
| Previously on SB204 at enrollment | xx (xx.x) |
| Completed Study | xx (xx.x) |
| SB204 Experienced | xx (xx.x) |
| SB204 Naïve | xx (xx.x) |
| Discontinued Early | xx (xx.x) |
| Primary Reason for Study Discontinuation [a] | |
| Adverse Events | xx (xx.x) |
| Lack of Efficacy as Determined by Investigator | xx (xx.x) |
| Withdrawal by Subject | xx (xx.x) |
| Physician Decision | xx (xx.x) |
| Protocol Violation | xx (xx.x) |
| Lost to Follow-up | xx (xx.x) |
| Pregnancy | xx (xx.x) |
| Worsening of Condition | xx (xx.x) |
| Other | xx (xx.x) |

Notes: Safety (SAF) Population includes all subjects that have been dispensed study drug and received at least one dose of SB204.

Unless stated otherwise, denominator is the number of subjects in safety population.

[a] Denominator is the number of subjects who were randomized.

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T xx.x x x xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Page x of y Novan Inc. Protocol Number: NI-AC303

Table 14.1.1.2 Summary of Protocol Deviations Safety Population

| Protocol Deviations | SB204<br>(N=XXX) |
|--------------------------------------|------------------|
| Subjects with Any Protocol Deviation | xxx (xx.x) |
| Deviation A | xxx (xx.x) |
| <br>Deviation B | xxx (xx.x) |
| <br>Deviation C | xxx (xx.x) |
| Etc. | |

Note (s): Percentages are based on the number of subjects in safety population. Reference: Listing 16.2.x

Protocol Number: NI-AC303

Table 14.1.2.1
Demographics
Safety Population

| | SB204 Experienced | SB204 Naïve | Overall |
|---|---|---|---|
| | (N=XXX) | (N=XXX) | (N=XXX) |
| Age (years) | | | |
| n | XXX | xxx | XXX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | X.X, XX.X | x.x, xx.x | x.x, xx.x |
| Age Group | | | |
| Juvenile (Age <18 years) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adult (Age 18+ years) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race | | | |
| White | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black or African American | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| American Indian or Alaska Native | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Native Hawaiian or Other Pacific | | | |
| Islander | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity | | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sex | | | |
| Male | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Female | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Previously in Study | | | |
| NI-AC301 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NI-AC302 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note(s): Percentages are based on the number of subjects in safety population. Age is based on the date of informed consent from the previous study (NI-AC301 or NI-AC302); LTS = Long Term Safety Study.

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T\_xx.x\_x\_x\_xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Novan Inc. Page x of y Protocol Number: NI-AC303

Table 14.1.2.2
Child Bearing Potential and Contraceptive Use (Females Only)
Safety Population

| | SB204 |
|----------------------------------------------------------------|-----------|
| | (N=XXX) |
| If Female, of Childbearing Potential? | |
| Yes | xx (xx.x) |
| No | xx (xx.x) |
| If No to Childbearing Potential, Why | |
| Post-Menopausal | xx (xx.x) |
| Hysterectomy or Bilateral Oophorectomy | xx (xx.x) |
| Surgically Sterilized | xx (xx.x) |
| If Yes to Childbearing Potential, Primary Method of Birth Cont | rol |
| Oral Contraceptive | xx (xx.x) |
| Intra-Uterine Device | xx (xx.x) |
| Condom with Spermicide | xx (xx.x) |
| Diaphragm with Spermicide | xx (xx.x) |
| Implant | xx (xx.x) |
| Nuvaring | xx (xx.x) |
| Medroxyprogesterone Injection | xx (xx.x) |
| Transdermal Patch | xx (xx.x) |
| Abstinence | xx (xx.x) |
| Other | xx (xx.x) |

Note(s): Percentages are based on the number of female subjects in Safety population. Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T xx.x x x xxxx.rtf, Generated on: DDMMMYYYY HH:MM Novan Inc. Page x of y Protocol Number: NI-AC303

Table 14.1.3

Medical History by System Organ Class and Preferred Term
Safety Population

| Body System Class | SB204 |
|---------------------------------------|-----------|
| Preferred Term | (N=XXX) |
| Subject with Any Medical History | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) |
| <br>Preferred Term n | xx (xx.x) |
| System Organ Class n | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) |
| <br>Preferred Term n | xx (xx.x) |
| | / |
| Sustan Organ Class a | xx (xx.x) |
| System Organ Class q Preferred Term 1 | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) |

Note(s): All investigator terms were coded using MedDRA dictionary version 18.1.

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T\_xx.x\_x\_x\_xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Protocol Number: NI-AC303

Table 14.1.4

Adverse Events Ongoing at the Start of the Study by System Organ Class, Preferred Term, and Extent of Exposure Safety Population

| System Organ Class<br>Preferred Term | SB204 Experienced (N=XXX) | SB204 Naïve<br>(N=XXX) | Overall (N=XXX) |
|---|---|---|---|
| Number of Subjects with at Least One Event | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Events | XX | XX | xx |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note(s): Adverse event terms were coded using MedDRA dictionary version 18.1. Subjects are counted once within each level of summary.

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T xx.x x x xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Programmer Note: Order SOC by decreasing frequency and preferred term by decreasing frequency within SOC based on overall incidence.

Protocol Number: NI-AC303

| Drug Class | SB204 |
|-------------------------------------------------------|-----------|
| Preferred Name | (N=XXX) |
| Subjects Who Took at Least One Concomitant Medication | xx (xx.x) |
| Drug Class 1 | xx (xx.x) |
| Preferred Name 1 | xx (xx.x) |
| Preferred Name 2 | xx (xx.x) |
| Preferred Name 3 | xx (xx.x) |
| etc. | xx (xx.x) |
| Drug Class 2 | xx (xx.x) |
| Preferred Name 1 | xx (xx.x) |
| Preferred Name 2 | xx (xx.x) |
| Preferred Name 3 | xx (xx.x) |
| etc. | xx (xx.x) |
| Drug Class 3 | xx (xx.x) |
| Preferred Name 1 | xx (xx.x) |
| Preferred Name 2 | xx (xx.x) |
| | xx (xx.x) |

Note(s): Subjects are counted only once at each level of summarization.

Concomitant medications are all medications taken during the study period, including those started before but ongoing at first dose. All medications were coded using WHO Drug dictionary version March 2016.

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T xx.x x x xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Programmer's Note(s): Continue with all drug classes and preferred names which appear in the data. Sort drug classes and within drug classes, preferred terms by decreasing overall frequency.

Protocol Number: NI-AC303

Table 14.2.1.

Summary of Duration and Extent of Drug Exposure
Safety Population

| | SB204 Experienced | SB204 Naïve | Overall |
|---|---|---|---|
| | (N=XXX) | (N=XXX) | (N=XXX) |
| Overall Duration of Exposure (Days) | | | |
| Number of Subjects with Exposure | xx | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | X.X, XX.X | X.X, XX.X | x.x, xx.x |
| Unknown | , | , | • |
| Days of Exposure | | | |
| n | xx | xx | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | X.X, XX.X | x.x, xx.x | X.X, XX.X |
| Unknown | | | |
| Areas of Application | | | |
| Face | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Upper Back | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Upper Chest | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Shoulders | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Extent of Exposure (grams) | | | |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | x.x, xx.x | x.x, xx.x | x.x, xx.x |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1-100 grams | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >100-330 grams | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >330-675 grams | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >675 grams | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Notes: All exposure endpoints includes exposure to SB204 from the previous study (NI-AC301 or NI-AC302), if applicable. Duration of Exposure = Date of Last Drug Administration - Date of First Drug Administration + 1 day. Days of exposure will be defined as the total number of days that the subject reported taking study medication. Areas of application indicate if the subject ever applied drug to that area. Each subject is counted only once per area.

Extent of exposure is determined as: 0.9 grams times the number of application areas times the number of days applied. Application to neck and jawline are considered part of application to the face when determining extent of exposure. Source: Listing xx.x.x.x.x, Program: xxxxx.sas, Output: T xx.x x x xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Protocol Number: NI-AC303

Table 14.2.2.1
Inflammatory Lesion Counts by Study Visit (Face Only)
Safety Population

| | | SB204<br>(N=XXX) | | |
|---|---|---|---|---|
| | | Count | Absolute Change | Percent Change |
| Visit | Statistic | | from Baseline | from Baseline |
| Baseline | N | XX | | |
| | Mean | XX.X | | |
| | SD | XX,XX | | |
| | Median | XX | | |
| | Min. to Max. | XX to XX | | |
| Week 4 | N | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX, XX | XX,XX | XX,XX |
| | Median | XX | XX,X | XX,X |
| | Min. to Max. | XX to XX | XX to XX | XX to XX |
| Week 12 | N | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X |
| | SD | XX,XX | XX,XX | XX,XX |
| | Median | XX | XX,X | XX,X |
| | Min. to Max. | XX to XX | XX to XX | XX to XX |

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T xx.x x x xxxx.rtf, Generated on: DDMMMYYYY HH:MM

### Programming Note: Repeat table for Non-Inflammatory Lesions:

Table 14.2.2.2 Non-Inflammatory Lesion Counts by Study Visit (Face Only) Safety Population

Protocol Number: NI-AC303

| _ | | SB204 Experienced (N=XXX) | | | SB204 Naïve<br>(N=XXX) | | |
|---|---|---|---|---|---|---|---|
| | · | Count | Absolute | Percent | Count | Absolute | Percent Change |
| | | | Change | Change | | Change | from Baseline |
| | | | from | from | | from | |
| Visit | Statistic | | Baseline | Baseline | | Baseline | |
| Baseline | N | XX | | | XX | | |
| | Mean | XX.X | | | XX.X | | |
| | SD | XX,XX | | | XX,XX | | |
| | Median | XX | | | XX | | |
| | Min. to Max. | XX to XX | | | XX to XX | | |
| Week 4 | N | XX | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX,XX | XX,XX | XX,XX | XX,XX | XX,XX | XX,XX |
| | Median | XX | XX,X | XX,X | XX | XX,X | XX,X |
| | Min. to Max. | XX to XX | XX to XX | XX to XX | XX to XX | XX to XX | XX to XX |
| Week 12 | N | XX | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX,XX | XX,XX | XX,XX | XX,XX | XX,XX | XX,XX |
| | Median | XX | XX,X | XX,X | XX | XX,X | XX,X |
| | Min. to Max. | XX to XX | XX to XX | XX to XX | XX to XX | XX to XX | XX to XX |

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T xx.x x x xxxx.rtf, Generated on: DDMMMYYYY HH:MM

### Programming Note: Repeat table for Non-Inflammatory Lesions:

Table 14.2.3.2 Non-Inflammatory Lesion Counts (Face Only) by Prior Treatment and Study Visit Safety Population

Protocol Number: NI-AC303

Table 14.3.1.1

Cutaneous Tolerability Evaluation - Erythema - Summarized by Study Visit (Face Only)

Safety Population

| | SB204 |
|--------------|-----------|
| Study Visit | (N=XXX) |
| Baseline | |
| 0 - None | xx (xx.x) |
| 1 - Mild | xx (xx.x) |
| 2 - Moderate | xx (xx.x) |
| 3 - Severe | xx (xx.x) |
| Missing | xx (xx.x) |
| Week 4 | |
| 0 - None | xx (xx.x) |
| 1 - Mild | xx (xx.x) |
| 2 - Moderate | xx (xx.x) |
| 3 - Severe | xx (xx.x) |
| Missing | xx (xx.x) |
| Week 12 | |
| 0 - None | xx (xx.x) |
| 1 - Mild | xx (xx.x) |
| 2 - Moderate | xx (xx.x) |
| 3 - Severe | xx (xx.x) |
| Missing | xx (xx.x) |
| Week 24 | |
| 0 - None | xx (xx.x) |
| 1 - Mild | xx (xx.x) |
| 2 - Moderate | xx (xx.x) |
| 3 - Severe | xx (xx.x) |
| Missing | xx (xx.x) |
| Week 36 | |
| 0 - None | xx (xx.x) |
| 1 - Mild | xx (xx.x) |
| 2 - Moderate | xx (xx.x) |
| 3 - Severe | xx (xx.x) |
| Missing | xx (xx.x) |
| Week 40\ET | |
| 0 - None | xx (xx.x) |
| 1 - Mild | xx (xx.x) |
| 2 - Moderate | xx (xx.x) |
| 3 - Severe | xx (xx.x) |
| Missing | xx (xx.x) |

Note: Baseline is the Week 12 assessment from the previous study (NI-AC301 or NI-AC302).

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T\_xx.x\_x\_x\_xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Protocol Number: NI-AC303

#### Using shell 14.3.1.1, repeat table for the following:

Table 14.3.1.2 Cutaneous Tolerability Evaluation - Scaling - Summarized by Study Visit Safety Population

Table 14.3.1.3 Cutaneous Tolerability Evaluation - Dryness - Summarized by Study Visit Safety Population

Table 14.3.1.4 Cutaneous Tolerability Evaluation - Pruritus - Summarized by Study Visit Safety Population

Table 14.3.1.5 Cutaneous Tolerability Evaluation - Burning/Stinging - Summarized by Study Visit Safety Population

Protocol Number: NI-AC303

Table 14.3.2.1

Shift from Baseline in Cutaneous Tolerability Evaluation - Erythema, by Study Visit (Face Only)

Safety Population

| Study Visit / | | Cutaneou | s Tolerability Score | at Baseline | |
|---|---|---|---|---|---|
| Cutaneous Tolerability | | | | | |
| Score | 0 - None | 1 - Mild | 2 - Moderate | 3 - Severe | Missing |
| 1 4 | | | | | |
| Week 4 | | | | | |
| 0 - None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 - Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 - Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 - Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 12 | | | | | |
| 0 - None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 - Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 - Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 - Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 24 | | | | | |
| 0 - None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 - Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 - Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 - Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 36 | | | | | |
| 0 - None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 - Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 - Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 - Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Week 40 | | | | | |
| 0 - None | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 - Mild | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 - Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 - Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Baseline is the Week 12 assessment from the previous study (NI-AC301 or NI-AC302).

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T\_xx.x\_x\_xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Protocol Number: NI-AC303

Using shell 14.3.2.1, Repeat table for the following:

Table 14.3.2.2 Shift from Baseline in Cutaneous Tolerability Evaluation - Scaling - Summarized Continuously by Study Visit Safety Population

Table 14.3.2.3 Shift from Baseline in Cutaneous Tolerability Evaluation - Dryness - Summarized Continuously by Study Visit Safety Population

Table 14.3.2.4 Shift from Baseline in Cutaneous Tolerability Evaluation - Pruritus - Summarized Continuously by Study Visit Safety Population

Table 14.3.2.5 Shift from Baseline in Cutaneous Tolerability Evaluation - Burning/Stinging - Summarized Continuously by Study Visit Safety Population

Protocol Number: NI-AC303

Table 14.3.3.1

Treatment Emergent Adverse Events (TEAE) Overview
Safety Population

| Number of Subjects with | SB204 Experienced (N=XXX) | SB204 Naïve<br>(N=XXX) | Overall (N=XXX) |
|---|---|---|---|
| Any TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of TEAEs | xx | xx | |
| Treatment-Related TEAE Number of Treatment-Related TEAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx | xx | xx |
| TEAE Leading to Treatment Modification | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of TEAE Leading to Treatment Modification | xx | xx | xx |
| Treatment-Related TEAE Leading to Treatment Modification Number of TRTEAE Leading to Treatment Modification | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx | xx | xx |
| TEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of TEAE Leading to Treatment Discontinuation | xx | xx | xx |
| Treatment-Related TEAE Leading to Treatment Discontinuation Number of TRTEAE Leading to Treatment Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx | xx | xx |
| Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Serious TEAEs | xx | xx | xx |
| Treatment-Related Serious TEAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Treatment-Related Serious TEAEs | xx | xx | xx |
| TEAE Leading to Death | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of TEAE Leading to Death | xx | xx | |
| Treatment-Related TEAE Leading to Death | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Treatment-Related TEAE Leading to Death | xx | xx | |

Note: TEAE onset is based on the start of treatment in the LTS. Adverse events were coded using MedDRA 18.1. TR=Treatment-Related.

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T\_xx.x\_x\_x\_x\_xxx.rtf, Generated on: DDMMMYYYY HH:MM

Protocol Number: NI-AC303

Table 14.3.3.2.1

Treatment Emergent Adverse Events (TEAE) by System Organ Class, Preferred Term, and Duration of Exposure Safety Population

| System Organ Class<br>Preferred Term | Within 24<br>hours<br>(N=XXX) | Within<br>2-30 days<br>(N=XXX) | Within<br>31-90<br>Days<br>(N=XXX) | Within<br>91-180<br>Days<br>(N=XXX) | Within<br>181-365<br>Days<br>(N=XXX) | Overall<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Number of Subjects with at Least One TEAE Number of Events | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x)<br>xx | xx (xx.x)<br>xx |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note(s): Adverse event terms were coded using MedDRA dictionary version 18.1. Subjects are counted once within each level of summary. Duration of exposure is based on date of first dose of SB204, which could be in the previous study (NI-AC301 or NI-AC302).

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T xx.x x x xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Programmer Note: Order SOC by decreasing frequency and preferred term by decreasing frequency within SOC based on overall incidence.

Protocol Number: NI-AC303

Table 14.3.3.2.2

Treatment Emergent Adverse Events (TEAE) by System Organ Class, Preferred Term, and Extent of Exposure Safety Population

| System Organ Class<br>Preferred Term | 1-100<br>grams<br>(N=XXX) | >100-330<br>grams<br>(N=XXX) | >330-675<br>grams<br>(N=XXX) | >675<br>Grams<br>(N=XXX) | Overall (N=XXX) |
|---|---|---|---|---|---|
| Number of Subjects with at Least One Event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of Events | xx | xx | xx | xx | xx |
| System Organ Class 1 Preferred Term 1 Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 2 Preferred Term 1 Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note(s): Adverse event terms were coded using MedDRA dictionary version 18.1. Subjects are counted once within each level of summary. TEAE onset is based on the start of treatment in the LTS. Extent of exposure is based on first exposure to SB204 - which could be in the previous study (NI-AC301 or NI-AC302).

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T xx.x x x xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Programmer Note: Order SOC by decreasing frequency and preferred term by decreasing frequency within SOC based on overall incidence.

Protocol Number: NI-AC303

#### Using shells 14.3.3.2.1 and 14.3.3.2.2, repeat for the following:

Table 14.3.3.3.1 Treatment-Related Emergent Adverse Events by System Organ Class, Preferred Term, and Duration of Exposure Safety Population

Table 14.3.3.3.2 Treatment-Related Emergent Adverse Events by System Organ Class, Preferred Term, and Extent of Exposure Safety Population

Programmer's Note: subset on TEAEs related to study treatment.

Table 14.3.3.4.1 Treatment Emergent Adverse Events Leading to Treatment Modification by Duration of Exposure Safety Population

Table 14.3.3.4.2 Treatment Emergent Adverse Events Leading to Treatment Modification by Extent of Exposure Safety Population

Programmer's Note: subset on TEAEs leading to treatment modification. Add the following footnote:

Note: Treatment modification includes reduction, interruption, or discontinuation of Study Drug

Table 14.3.3.5.1 Treatment-Related Treatment Emergent Adverse Events Leading to Treatment Modification by Duration of Exposure Safety Population

Table 14.3.3.5.2 Treatment-Related Treatment Emergent Adverse Events Leading to Treatment Modification by Extent of Exposure Safety Population

Programmer's Note: subset on Treatment-Related TEAEs leading to treatment modification. Add the following footnote:

Note: Treatment modification includes reduction, interruption, or discontinuation of Study Drug.

Table 14.3.3.6.1 Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug by Duration of Exposure Safety Population

Table 14.3.3.6.2 Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug by Extent of Exposure Safety Population

Programmer's Note: subset on TEAEs leading to discontinuation of Study Drug.

Table 14.3.3.7.1 Treatment-Related Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug by Duration of Exposure Safety Population

Protocol Number: NI-AC303

Table 14.3.3.7.2 Treatment-Related Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug by Extent of Exposure Safety Population

Programmer's Note: subset on Treatment-Related TEAEs leading to discontinuation of Study Drug.

Table 14.3.3.8.1 Treatment Emergent Serious Adverse Events by System Organ Class, Preferred Term, and Duration of Exposure Safety Population

Table 14.3.3.8.2 Treatment Emergent Serious Adverse Events by System Organ Class, Preferred Term, and Extent of Exposure Safety Population

Programmer's Note: subset on Serious TEAEs.

Table 14.3.3.9.1 Treatment-Related Treatment Emergent Serious Adverse Events by System Organ Class, Preferred Term, and Duration of Exposure Safety Population

Table 14.3.3.9.2 Treatment-Related Treatment Emergent Serious Adverse Events by System Organ Class, Preferred Term, and Extent of Exposure Safety Population

Programmer's Note: subset on Treatment-Related Serious TEAEs.

Table 14.3.3.10.1 Treatment Emergent Adverse Events Leading to Death by Duration of Exposure Safety Population Table 14.3.3.10.2 Treatment Emergent Adverse Events Leading to Death by Extent of Exposure Safety Population

Programmer's Note: subset on TEAEs with fatal outcome.

Table 14.3.3.11.1 Treatment-Related Treatment Emergent Adverse Events Leading to Death by Duration of Exposure Safety Population

Table 14.3.3.11.2 Treatment-Related Treatment Emergent Adverse Events Leading to Death by Extent of Exposure Safety Population

Programmer's Note: subset on treatment related TEAEs with fatal outcome.

•

Protocol Number: NI-AC303

Table 14.3.3.13

Summary of Treatment Emergent Adverse Events (TEAE) by Highest Severity, System Organ Class and Preferred Term Safety Population

| System Organ Class | | SB204 |
|----------------------------------|----------|-----------|
| Preferred Term | Severity | (N=XXX) |
| Subjects with at least one event | Mild | xx (xx.x) |
| | Moderate | xx (xx.x) |
| | Severe | xx (xx.x) |
| Number of events | Mild | XX |
| | Moderate | XX |
| | Severe | XX |
| System Organ Class 1 | Mild | xx (xx.x) |
| | Moderate | xx (xx.x) |
| | Severe | xx (xx.x) |
| Preferred Term 1 | Mild | xx (xx.x) |
| | Moderate | xx (xx.x) |
| | Severe | xx (xx.x) |

Note(s): TEAE onset is based on the start of treatment in the LTS. Adverse event terms were coded using MedDRA dictionary version 18.1. Subjects are counted once within each level of summary. If a subject has multiple events, the event with highest severity will be considered.

Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T xx.x x x xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Programmer Note: Order SOC by decreasing frequency and preferred term by decreasing frequency within SOC based on overall incidence.

Protocol Number: NI-AC303

#### Using shell 14.3.3.13, repeat table for the following:

Table 14.3.3.14 Summary of Treatment-Related Emergent Adverse Events (TEAE) by Severity, System Organ Class and Preferred Term Safety Population

Programmer's Note: subset on related TEAEs

Protocol Number: NI-AC303

Table 14.3.4
Summary of Vital Signs
Safety Population

#### <Parameter> (<units>)

| | - | SB204 |
|-----------|--------------|----------------------|
| | | N=XXX) |
| Timepoint | Actual | Change from Baseline |
| Baseline | | |
| n | XX | |
| Mean (SD) | xx.x (xx.xx) | |
| Median | XX.X | |
| Min, Max | XX, XX | |
| Missing | xx | |
| Week 4 | | |
| N | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX |
| Missing | xx | XX |
| Week 12 | | |
| n | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx |
| • • • • | | XX |

Note(s): Baseline is defined as the Week 12 assessment from the previous study (NI-AC301 or NI-AC302). Source: Listing xx.x.x.x, Program: xxxxx.sas, Output: T\_xx.x\_x\_x\_xxxx.rtf, Generated on: DDMMMYYYY HH:MM

Programmer Note: Include all vital signs parameters (e.g. SBP, DBP, Pulse) and all available post-baseline visits. Missing not presented if no missing values.
#### **Protocol: NI-AC303**

A Phase 3 Multi-Center, Open Label Study Evaluating the Long Term Safety of SB204 Once Daily in the Treatment of Acne Vulgaris.

Mock Data Displays - Figures Version 1.0 Date: 12Apr2017

> Prepared for: Novan Inc. 4105 Hopson Road Morrisville, NC 27560

Prepared by:
Chiltern International
4000 CentreGreen Way, Suite 300, Cary, NC, 27513, United States

This document is the confidential information of Novan Inc. It may not be disclosed to parties not associated with the clinical investigation or used for any purpose without the prior written consent of Novan Inc.

Contents

| Figure 14.1.1 Distribution of Erythema Scores by Treatment and Visit Safety Population |
|---|
| Figure 14.1.2 Distribution of Dryness Scores by Treatment and Visit, Safety Population |
| Figure 14.1.3 Distribution of Scaling Scores by Treatment and Visit, Safety Population |
| Figure 14.1.4 Distribution of Pruritus Scores by Treatment and Visit, Safety Population |
| Figure 14.1.5 Distribution of Burning/stinging Scores by Treatment and Visit, Safety Population |
| Figure 14.2.1 Average Change from Baseline in Inflammatory Lesion Count Over Time Safety Population |
| Figure 14.2.2 Average Percent Change from Baseline in Inflammatory Lesion Count Over Time Safety Population |
| Figure 14.3.1 Average Change from Baseline in Non-Inflammatory Lesion Count Over Time, Safety Population7 |
| Figure 14.3.2 Average Percent Change from Baseline in Non-Inflammatory Lesion Count Over Time, Safety Population 7 |

Figure 14.1.1 Distribution of Erythema Scores by Treatment and Visit Safety Population

Figure 14.1.1
Distribution of Erythema Scores by Treatment and Visit
Safety Population



Using shell for Figure 14.1.1, repeat for the following:

Figure 14.1.2 Distribution of Dryness Scores by Treatment and Visit, Safety Population

Figure 14.1.3 Distribution of Scaling Scores by Treatment and Visit, Safety Population

Figure 14.1.4 Distribution of Pruritus Scores by Treatment and Visit, Safety Population

Figure 14.1.5 Distribution of Burning/stinging Scores by Treatment and Visit, Safety Population

Figure 14.2.1 Average Change from Baseline in Inflammatory Lesion Count (Face only) Over Time Safety Population

 $\begin{tabular}{lll} Figure 14.2.1 \\ Average Change from Baseline in Inflammatory Lesion Count Over Time \\ Safety Population \\ \end{tabular}$ 



Figure 14.2.2 Average Percent Change from Baseline in Inflammatory Lesion Count (Face only) Over Time
Safety Population

Figure 14.2.2

Average Percent Change from Baseline in Inflammatory Lesion Count Over Time
Safety Population



Using shell for Figure 14.2.1, repeat for the following:

Figure 14.3.1 Average Change from Baseline in Non-Inflammatory Lesion Count (Face only) Over Time, Safety Population

Using shell for Figure 14.2.2 repeat for the following:

Figure 14.3.2 Average Percent Change from Baseline in Non-Inflammatory Lesion Count (Face only) Over Time, Safety Population

**Protocol: NI-AC303** 

A Phase 3 Multi-Center, Open Label Study Evaluating the Long Term Safety of SB204 Once Daily in the Treatment of Acne Vulgaris.

Mock Data Displays- Listings Version 1.0 Date: 12Apr2017

> Prepared for: Novan Inc. 4105 Hopson Road Morrisville, NC 27560

Prepared by: Chiltern International 4000 CentreGreen Way, Suite 300, Cary, NC, 27513, United States

This document is the confidential information of Novan Inc. It may not be disclosed to parties not associated with the clinical investigation or used for any purpose without the prior written consent of Novan Inc.

#### **Table of Contents**

| Listing 16.2.1.1 Subject Disposition Safety Population | 3 |
|---|---|
| Listing 16.2.1.1 Subject Disposition Safety Population Listing 16.2.2 Protocol Violations/Deviations Safety Population Listing 16.2.3 Inclusion/Exclusion Criteria not Met Safety Population | 4 |
| Listing 16.2.3 Inclusion/Exclusion Criteria not Met Safety Population | 5 |
| Listing 16.2.4.1 Demographics Safety Population | 6 |
| Listing 16.2.4.2 Medical History Safety Population | 7 |
| Listing 16.2.4.3 Child Bearing Potential and Pregnancy Test Results Safety Population (Females only) | 8 |
| Listing 16.2.4.4 Physical Exam Safety Population | 9 |
| Listing 16.2.5 Study Drug Management Safety Population | |
| Listing 16.2.6 Extent and Duration of Exposure Safety Population | 11 |
| Listing 16.2.7.1.1 Lesion Counts: Total Inflammatory and Non-Inflammatory Lesions Safety Population | 12 |
| Listing 16.2.7.1.2 Lesion Counts: Papules, Pustules, Nodules, and Cysts Safety Population | 13 |
| Listing 16.2.7.3 Cutaneous Tolerability Safety Population | 14 |
| Listing 16.2.7.4 Vital Signs Safety Population | 15 |
| Listing 16.2.7.5 Concomitant Medications Safety Population | 16 |
| Listing 16.2.8.1 Adverse Events Safety Population | 17 |
| Listing 16.2.8.2 Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug Safety Population | 18 |
| Listing 16.2.8.3 Treatment-Emergent Adverse Events Leading to Treatment Modification Safety Population | 18 |
| Listing 16.2.8.4 Treatment-Emergent Serious Adverse Events Safety Population | 18 |
| Listing 16.2.8.5 Treatment-Emergent Adverse Events Leading to Death Safety Population | 18 |
| Listing 16.2.9 Concomitant Medical and Surgical Procedures Safety Population | 19 |

Novan Inc
Protocol Number: NI-AC303

Listing 16.2.1.1

| ттасти | g 10.2.1.1 |
|---------|-------------|
| Subject | Disposition |
| Safety | Population |

| Previous<br>Study | Previous<br>Treatment<br>Group | Subject<br>ID | Met All<br>Inc/Exc<br>Criteria | Date of:<br>Informed<br>Consent | Date of<br>Completion or<br>Discontinuation | Reason for Discontinuation |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | xxxxxxx | Yes | DDMMMYYYY | DDMMMYYYY | Completed |
| xxxxxxxx | xxxxxxx | xxxxxxxx | Yes | DDMMMYYYY | DDMMMYYYY | Withdrawal by Subject |

s<nnn>xxxx yyyymmddthh:mm

Programmer's Note(s): This listing will be sorted by previous study number and then by Subject ID.

Protocol Number: NI-AC303

### Listing 16.2.2 Protocol Violations/Deviations Safety Population

| Subject ID | Date of<br>Violation/<br>Deviation<br>/Day | Type of Violation | Details of Violation/Deviation |
|---|---|---|---|
| xxxxxx | DDMMMYYYY/xx | ICF Issue | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxxx | DDMMMYYYY/xx | Assessment not<br>Performed per Protocol | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxxx | DDMMMYYYY/xx | Non-compliance with IP | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Note(s): Day = Day relative to the date of first dose of study medication. s<nnn>xxxx yyyymmddthh:mm

Programmer's Note(s): This and subsequent listings will be sorted by Subject ID.

Protocol Number: NI-AC303

# Listing 16.2.3 Inclusion/Exclusion Criteria not Met Safety Population

| Subject ID | Criteria Not Met | Description of Criteria |
|------------|------------------|-------------------------|
| xxxxxx | INCXX | xxxxxxxxxxxxxxxxx |
| XXXXXXX | EXCLXX | xxxxxxxxxxxxxxxxx |

Protocol Number: NI-AC303

Listing 16.2.4.1
Demographics
Safety Population

| Subject ID | Study<br>Center | Date of<br>Birth | Age<br>(years) | Gender | Ethnicity | Race |
|---|---|---|---|---|---|---|
| xxxxxxx | xxxxxxx | DDMMMYYYY | XX.X | Male | Not Hispanic or<br>Latino | xxxxxx |
| xxxxxxx | xxxxxx | DDMMMYYYY | xx.x | Female | Not Hispanic or<br>Latino | xxxxx |
| xxxxxxx | xxxxxx | DDMMMYYYY | XX.X | Female | Not Hispanic or<br>Latino | Other: xxxxxx |

Note(s): Age is calculated as the interval between date of birth and date of baseline visit from the previous study (NI-AC301 or NI-AC302).

s<nnn>xxxx yyyymmddthh:mm

Protocol Number: NI-AC303

Listing 16.2.4.2 Medical History Safety Population

| Subject ID | SOC /<br>Preferred Term /<br>Verbatim Term | Onset / End |
|---|---|---|
| xxxxxx | Xxxxxxxx /<br>Xxxxxxxx /<br>xxxxxxxx | DDMMYYYY / DDMMYYYY |
| xxxxxxx | Xxxxxxx /<br>Xxxxxxxx /<br>xxxxxxxx | DDMMYYYY / Ongoing |

s<nnn>xxxx yyyymmddthh:mm

Protocol Number: NI-AC303

# Listing 16.2.4.3 Child Bearing Potential and Pregnancy Test Results Safety Population (Females only)

| Subject ID | Of Child-<br>Bearing<br>Potential? | If no, why? | If Yes, Method<br>of Birth Control | Visit | Collection Date<br>/ Day | Pregnancy Test<br>Result or<br>Reason Not Done |
|---|---|---|---|---|---|---|
| XXXXXXX | Yes<br>No | XXXXXXXXXXX | xxxxxxxxx | Baseline<br>Baseline | DDMMMYYYY /XX<br>DDMMMYYYY /XX | Negative<br>Negative |

Note(s): Day = Day relative to the date of first day of LTS. s<nnn>xxxx yyyymmddthh:mm

Novan Inc
Protocol Number: NI-AC303

Safety Population

Listing 16.2.4.4
Physical Exam

| Subject ID | Visit | Date | Body System | Evaluation | Abnormality |
|---|---|---|---|---|---|
| XXXXXXX | Baseline | DDMMMYYYY | General Appearance<br>Respiratory<br>Cardiovascular<br>Other: XXXXXXXX | Normal<br>Normal<br>Normal<br>ANCS | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | Week 40\ET | DDMMMYYYY | General Appearance Respiratory Cardiovascular | ACS Normal | xxxxxxxxxxxxxxx |
| | Etc. | | cararovascurar | NOTHIAL | |
| XXXXXXX | Baseline | DDMMMYYYY | General Appearance<br>Respiratory | Normal<br>Normal | |

Note(s):ANCS = Abnormal, Not clinically significant; ACS = Abnormal, Clinically Significant. If a finding was determined to be clinically significant, it is also reported as an adverse event, or, if it occurred prior to study start, it is reported in medical history. s<nnn>xxxx yyyymmddthh:mm

Protocol Number: NI-AC303

Listing 16.2.5
Study Drug Management
Safety Population

| Subject | | | Was Pump | | | Was previous | |
|---|---|---|---|---|---|---|---|
| ID | Visit | Date/ Day | dispensed? | If yes, | Pump number(s) | pump returned? | If no. Reason why: |
| | | , | | | | | |
| XXXXXXX | Baseline | DDMMMYYYY/xx | Yes | XXXXXX | | | |
| | Week 4 | DDMMMYYYY/xx | No | | | No | XXXXXXXXX |
| | Week 12 | DDMMMYYYY/xx | Yes | XXXXXX, | XXXXX | | |
| | Week 24 | DDMMMYYYY/xx | Yes | XXXXXX, | XXXXX, XXXXX | | |
| | Week 36 | DDMMMYYYY/xx | Yes | XXXXXX | | | |
| | Week 40 | DDMMMYYYY/xx | Yes | XXXXXX | | | |
| Xxxxxxx | Baseline | DDMMMYYYY/xx | Yes | XXXXXX | | | |
| | Week 4 | DDMMMYYYY/xx | Yes | XXXXXX | | | |
| | Week 12 | DDMMMYYYY/xx | Yes | XXXXXX | | Yes | |
| | Week 24 | DDMMMYYYY/xx | Yes | XXXXXX | | | |
| | Week 36 | DDMMMYYYY/xx | Yes | XXXXXX | | | |
| | Week 40 | DDMMMYYYY/xx | Yes | XXXXXX | | | |
| xxxxxxx | Baseline | DDMMMYYYY/xx | Yes | XXXXXX | | | |
| *************************************** | Week 4 | DDMMMYYYY/xx | Yes | XXXXXX | | Yes | |
| | Week 12 | DDMMMYYYY/xx | Yes | XXXXXX | | 105 | |
| | Week 24 | DDMMMYYYY/xx | No | | | | |
| | Week 36 | DDMMMYYYY/xx | Yes | XXXXXX | | | |
| | Week 40 | DDMMMYYYY/xx | Yes | XXXXXX | | | |
| | WCCI 40 | DDIMMITTIT/ AA | 100 | 2121212121 | | | |

Note(s): Day = Day relative to the date of first day of LTS.

Protocol Number: NI-AC303

Listing 16.2.6
Extent and Duration of Exposure
Safety Population

| Subject<br>ID | Visit | Date | Duration<br>of<br>Exposure<br>(days) | Number of<br>Doses<br>Reported<br>Missed | | | | | | Areas | of Applicat | ion |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Days of<br>Exposure | of<br>Exposure<br>(grams) | Face | Upper<br>Back | Upper<br>Chest | Shoulders | Other: | |
| | 57 - 1 4 | | 77777 | 373737 | 77777 | 171717 | | ** | | | | |
| XXXXXXX | Week 4 | DDMMMYYYY | XXX | XXX | XXX | XXX | X | X | | | | |
| | Week 12 | DDMMMYYYY | XXX | XXX | XXX | XXX | | X | | X | | |
| | Week 24 | DDMMMYYYY | XXX | XXX | XXX | XXX | | | X | X | | |
| | Week 36 | DDMMMYYYY | UNK | UNK | UNK | UNK | | | | X | Neck and Jawline | |
| | Week 40 | DDMMMYYYY | XXX | XXX | XXX | XXX | | | | | | |
| | Overall | | XXX | UNK | UNK | UNK | | | | | | |
| | | | | | | | | | | х | xxxxxxxxx | |
| Xxxxxx | Week 4 | DDMMMYYYY | XXX | XXX | XXX | XXX | | | | | | |
| | Week 12 | DDMMMYYYY | XXX | XXX | XXX | XXX | | | | | | |
| | Week 24 | DDMMMYYYY | XXX | XXX | XXX | XXX | | | | | | |
| | Week 36 | DDMMMYYYY | XXX | XXX | XXX | XXX | | | | | | |
| | Week 40 | DDMMMYYYY | XXX | XXX | XXX | XXX | | | | | | |
| | Overall | | XXX | XXX | XXX | XXX | | | | | | |

#### Note(s):

Duration of Exposure = (Date of next drug dispensation or if last dispensataion, date of last dose) - Date of Drug Dispensation + 1 day. Overall is based on the date of first dose of study drug, which could be from the previous study (NI-AC301 or NI-AC302).

Days of Exposure = Duration of exposure minus the number of days that the subject reported not taking study medication. Extent of Exposure: Each application is equal to 0.9 g. Extent of exposure is estimated as the sum of application areas (face only=1, face and chest=2, etc) times the number of days of application to those areas times 0.9g. If the other specification is jaw or neckline, it is assumed that the same pump stroke used to apply drug to face is being used for the jaw and/or neckline application. For subjects randomized to SB204 in the previous studies, drug was only applied to the face so for the days of exposure from the previous studies, it will be assumed that there is only one area of application, i.e. the face.

UNK = Unknown: For subjects who are lost-to-follow-up or who did not return diaries but reported an unknown number of missed doses, duration of exposure and days of exposure for that visit interval are defined as unknown. Overall duration will be defined as above; days of exposure will remain unknown.

Protocol Number: NI-AC303

Listing 16.2.7.1.1

Lesion Counts (Face Only): Total Inflammatory and Non-Inflammatory Lesions
Safety Population

| | | | | _ | Infl | Lammatory Le | sions | Non-Ir | nflammatory : | Lesions |
|---|---|---|---|---|---|---|---|---|---|---|
| Previous | Subject | | | Counter's | | Absolute<br>Change<br>from | Percent<br>Change<br>from | | Absolute<br>Change<br>from | Percent<br>Change<br>from |
| Study | ID | Visit | Date | Initials | Count | Baseline | Baseline | Count | Baseline | Baselin |
| | | Baseline | DDMMMYYYY | XXXX | XX | | | XX | | |
| XXXXXX | XXXXXXX | Week 4 | DDMMMYYYY | XXXX | XX | XX | XX | XX | XX | XX |
| | | | | | XX | XX | XX | XX | XX | XX |
| | | Week 12 | DDMMMYYYY | XXXX | | | | | | |
| | | Week 24 | DDMMMYYYY | XXXX | XX | XX | XX | XX | XX | XX |
| | | Week 36 | DDMMMYYYY | XXXX | XX | XX | XX | XX | XX | XX |
| | | Week 40 | DDMMMYYYY | XXXX | XX | XX | XX | XX | XX | XX |
| xxxxxx | xxxxxxx | Baseline | DDMMMYYYY | XXXX | XX | | | XX | | |
| | | Week 4 | DDMMMYYYY | XXXX | XX | XX | XX | XX | XX | XX |
| | | Week 12 | DDMMMYYYY | XXXX | XX | XX | XX | XX | XX | XX |
| | | Week 24 | DDMMMYYYY | XXXX | XX | XX | XX | XX | XX | XX |
| | | Week 36 | DDMMMYYYY | XXXX | XX | XX | XX | XX | XX | XX |
| | | Week 40 | DDMMMYYYY | XXXX | XX | XX | XX | XX | XX | XX |

Note: Inflammatory Lesions includes: papules/pustules + nodules/cysts.s<nnn>xxxx yyyymmddthh:mm

Novan Inc
Protocol Number: NI-AC303

Listing 16.2.7.1.2

Lesion Counts (Face Only): Papules, Pustules, Nodules, and Cysts

Safety Population

| Previous Study | Subject ID | Visit | Date | Counter's<br>Initials | Papules/Pustules | Nodules/Cyst: |
|---|---|---|---|---|---|---|
| rievieus seud <sub>i</sub> | 542,555 12 | 11010 | 2400 | 111101010 | rapares, rassares | reaures, e <sub>1</sub> s e. |
| xxxxxx | xxxxxxx | Baseline | DDMMMYYYY | XXXX | XXX | XXX |
| | | Week 4 | DDMMMYYYY | XXXX | XXX | XXX |
| | | Week 12 | DDMMMYYYY | XXXX | XXX | XXX |
| | | Week 24 | DDMMMYYYY | XXXX | XXX | XXX |
| | | Week 36 | DDMMMYYYY | XXXX | XXX | XXX |
| | | Week 40 | DDMMMYYYY | XXXX | XXX | XXX |
| xxxxxx | xxxxxx | Baseline | DDMMMYYYY | XXXX | XXX | XXX |
| | | Week 4 | DDMMMYYYY | XXXX | XXX | XXX |
| | | Week 12 | DDMMMYYYY | XXXX | XXX | XXX |
| | | Week 24 | DDMMMYYYY | XXXX | XXX | XXX |
| | | Week 36 | DDMMMYYYY | XXXX | XXX | XXX |
| | | Week 40 | DDMMMYYYY | XXXX | XXX | XXX |

Protocol Number: NI-AC303

Listing 16.2.7.3 Cutaneous Tolerability Safety Population

| Previous<br>Study | Subject<br>ID | Visit | Date | Erythema | Scaling | Dryness | Pruritus | Burning/<br>Stinging |
|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xxxxxxx | Baseline | DDMMMYYYY | Mild | Mild | Moderate | None | None |
| | | Week 4 | DDMMMYYYY | Mild | Mild | Moderate | None | None |
| | | Week 12 | DDMMMYYYY | Mild | Mild | Moderate | None | None |
| | | Week 24 | DDMMMYYYY | Mild | Mild | Moderate | None | None |
| | | Week 36 | DDMMMYYYY | Mild | Mild | Moderate | None | None |
| | | Week 40 | DDMMMYYYY | Mild | Mild | Moderate | None | None |
| xxxxxxx | xxxxxxxx | Baseline | DDMMMYYYY | Mild | Mild | Moderate | None | None |
| | | Week 4 | DDMMMYYYY | Mild | Mild | Moderate | None | None |
| | | Week 12 | DDMMMYYYY | Mild | Mild | Moderate | None | None |
| | | Week 24 | DDMMMYYYY | Mild | Mild | Moderate | None | None |
| | | Week 36 | DDMMMYYYY | Mild | Mild | Moderate | None | None |
| | | Week 40 | DDMMMYYYY | Mild | Mild | Moderate | None | None |

Note(s): 0 = None, 1 = Mild, 2=Moderate, 3 = Severe. s<nnn>xxxx yyyymmddthh:mm

Protocol Number: NI-AC303

Listing 16.2.7.4 Vital Signs Safety Population

| Previous<br>Study | Subject ID | Visit | Date/ Day | Systolic<br>BP (mmHg) | Diastolic<br>BP (mmHg) | Pulse<br>(bpm) | Evaluation | If Abnormal and<br>Clinically<br>Significant, provide<br>MH or AE term |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | Baseline | DDMMMYYYY/xx | xxx | xxx | XXX | Normal | |
| | | Week 4 | DDMMMYYYY/xx | XXX | XXX | XXX | Abnormal, NCS | |
| | | Week 12 | DDMMMYYYY/xx | XXX | XXX | XXX | Normal | |
| | | Week 24 | DDMMMYYYY/xx | XXX | XXX | XXX | Normal | |
| | | Week 36 | DDMMMYYYY/xx | XXX | XXX | XXX | Normal | |
| | | Week 40 | DDMMMYYYY/xx | XXX | XXX | xxx | Normal | |
| xxxxxxx | xxxxxxx | Baseline | DDMMMYYYY/xx | xxx | xxx | xxx | Abnormal, CS | xxxxxxxxxxx |

Note(s): Day = Day relative to the first day of LTS. NCS = Not clinically significant; CS = Clinically Significant. If a post-baseline finding was determined to be clinically significant, it is also reported as an adverse event. s<nnn>xxxx yyyymmddthh:mm Novan Inc
Protocol Number: NI-AC303

Listing 16.2.7.5

| Listing 16.2./.5 |
|-------------------------|
| Concomitant Medications |
| Safety Population |

| Previous<br>Study | Subject ID | Drug Class/<br>Preferred Name/<br>Reported Term | Indication | Start Date (Day)/<br>End Date (Day) | Dose (Unit) /<br>Frequency /<br>Route | If for AE or<br>MH, Primary<br>Term | Ongoing from<br>Previous<br>Study? |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXX/<br>XXXXXXX | Adverse Event | DDMMMYYYY (XX)/<br>Ongoing | | | |
| xxxxxxx | xxxxxxx | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | Medical History | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | XXX.X (XXXXX) / XXX / XXXXXXXXX | XXXXXXXX | Yes |
| xxxxxx | xxxxxx | xxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxxx | Prophylaxis | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | XXX.X (XXXXX) / XXX / XXXXXXXXX | | |
| xxxxxxx | xxxxxxx | xxxxxxxxxxxx/<br>xxxxxxxxxxxxx/<br>xxxxxxxxxx | Dietary Supplement | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | XXX.X (XXXXX) / XXX / XXXXXXXXX | XXXXXXXX | No |
| xxxxxxx | xxxxxxx | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxx/<br>xxxxxxxx | Contraception | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | XXX.X (XXXXX) /<br>XXX /<br>XXXXXXXXX | | |
| xxxxxxx | xxxxxxx | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXXX | Other: XXXXXXXXXXX | DDMMMYYYY (XX)/<br>DDMMMYYYY (XX) | XXX.X (XXXXX) / XXX / XXXXXXXXX | | |

Note(s): Day = Day relative to the first day of LTS. Coding will be done using the WHO March 2016 dictionary. Drug Class corresponds to ACT level 2. s<nnn>xxxx yyyymmddthh:mm

Protocol Number: NI-AC303

Listing 16.2.8.1
Adverse Events
Safety Population

| Subject ID | Duration<br>of<br>Exposure<br>(days) | Extent<br>of<br>Exposure<br>(grams) | System Organ Class/<br>Preferred Term/<br>Reported Term | T<br>E<br>A<br>E | First Dose Date/ Start Date/ End Date / (Days) | Cause<br>Study<br>Discon-<br>tinuation? | Severity /<br>Relationship | Action /<br>Treatment /<br>Final<br>Outcome | SAE? | SAE<br>Criteria |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xx | xx.x | XXXXXXXXXXXXXXX /<br>XXXXXXXXXXXXX /<br>XXXXXXXX | Y | DDMMMYYY /<br>DDMMMYYYY /<br>DDMMMYYYY /<br>XX | No | Mild /<br>Unlikely | Dose Not<br>Changed /<br>XXXXXXXX /<br>XXXXXXXXXXXXXXX | No | |
| xxxxxx | XX | XX.X | XXXXXXXXXXXXXX /<br>XXXXXXXXXXXXX /<br>XXXXXXXX | Y | DDMMMYYY /<br>DDMMMYYY /<br>DDMMMYYYY /<br>XX | Yes | XXXXXXX /<br>XXXXXXX | XXXXXXXXX /<br>XXXXXXXXX /<br>XXXXXXXXXXXXXXX | Yes | XXXXXXXXX<br>XX |

Note(s): TEAE=Treatment-emergent Adverse Event. TEAE onset is based on the start of treatment in the LTS. Days = (Adverse event end date - event start date)+1. Adverse events were coded using MedDRA 18.1. Duration and extent of exposure are based on the date of first dose of study drug, which could from the previous study (NI-AC301 or NI-AC302). s<nnn>xxxx yyyymmddthh:mm

Protocol Number: NI-AC303

Repeat Listing 16.2.8.1 for:

Listing 16.2.8.2 Treatment-Emergent Adverse Events Leading to Discontinuation of Study Drug Safety Population

Listing 16.2.8.3 Treatment-Emergent Adverse Events Leading to Treatment Modification Safety Population

Listing 16.2.8.4 Treatment-Emergent Serious Adverse Events Safety Population

Listing 16.2.8.5 Treatment-Emergent Adverse Events Leading to Death Safety Population

Protocol Number: NI-AC303

Listing 16.2.9 Concomitant Medical and Surgical Procedures Safety Population

| Previous<br>Study | Subject ID | Verbatim Term | Start Date (Day) /<br>End Date (Day) | Was it for an AE/SAE? | Ongoing from<br>Previous<br>Study? |
|---|---|---|---|---|---|
| xxxxxx | xxxxxx | xxxxxxxxxxxxxxxx | DDMMYYYY (XX) /<br>DDMMYYYY (XX) | No | Yes |
| xxxxxxx | xxxxxxx | xxxxxxxxxxxxxxxxx | DDMMYYYY (XX) /<br>Ongoing | No | No |